CLINICAL TRIAL: NCT01499537
Title: Prospective Randomized Study of PTC and EUS-guided Drainage of the Bile Duct in Patients With Malignant or Post-operative Jaundice After Failure or Impossibility to Perform Endoscopic Retrograde Cholangiography
Brief Title: Prospective Randomized Study of PTC and EUS-guided Drainage of the Bile Duct
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHAGE/IPC 2010-002
Record Dates: First submitted 2011-09-16; First posted 2011-12-26 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-02

CONDITIONS: Jaundice
Keywords: Stenosis of biliary ways
MeSH Terms: conditions — Jaundice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Percutaneous Drainage (Active Comparator): Percutaneous Transhepatic Biliary Drainage (PTBD)
  Interventions: Device: biliary drainage
- EUS-guided drainage (Experimental): endoscopic ultrasonography guided biliary drainage through the duodenal or the gastric wall
  Interventions: Device: EUS guided biliary drainage

INTERVENTIONS:
Device: biliary drainage — percutaneous transhepatic biliary drainage (PTBD)
  Arms: Percutaneous Drainage
Device: EUS guided biliary drainage — endoscopic ultrasonography guided biliary drainage through the duodenal or the gastric wall
  Arms: EUS-guided drainage

SUMMARY:
At this time, endoscopic retrograde cholangiopancreatography (ERCP) stay the gold standard method to achieve biliary drainage in case of malignant or benign stricture. When ERCP fail or if the major papilla is not suitable, percutaneous transhepatic biliary drainage (PTBD) is the most commonly used alternative, surgery having higher morbidity and mortality rates, unacceptable especially in palliative situation. Recent developments in interventional endoscopic ultrasonography (EUS) allow new endoluminal approaches to pancreatic-biliary structures, such as cysto-enterostomy or pancreatic-enterostomy. More recently were described the possibility to realize EUS-guided biliary drainage, through the duodenal or the gastric wall. Advantages of the EUS-guided approach are to be realizable even the papilla is not suitable endoscopically (duodenal stricture or post-surgical status) and to allow if necessary extra-tumoral non anatomic drainage (hepaticogastrostomy). This technique is actually an alternative to PTBD. In comparison of the PTBD, EUS-guided route seems to have less morbidity and to avoid external biliary drainage. Indeed, the morbidity rate of the percutaneous biliary drainage and the EUS-guided biliary drainage range respectively from 25 to 35% and from 0 to 23%. However, none study compare prospectively both techniques. Aims of this study are to compare the morbidity rate, feasibility and efficacy of these techniques.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18
* Karnofsky >= 50%
* biliary stenosis (malignant or benign stricture)with failure of endoscopic retrograde cholangiopancreatography
* signed informed consent

Exclusion Criteria:

* isolated biliary stenosis of right hepatic canal
* percutaneous biliary drainage < 10 days
* laparotomy < 10 days
* contra-indication to the procedure
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-01; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Morbidity rate | 30 days
  Morbidity rate during 30 post-operative days

SECONDARY OUTCOMES:
efficacy | 15 days
  decrease of bilirubine > 50%
feasibility | up to 3 days
  succes or not of the intervention to obtain bilairy drainage
biliary drainage duration | up to 1 month
  time between intervention and drain withdrawal
quality of life | 30 days
  QLQ-C30 questionnary at inclusion and at D30

CONTACTS AND LOCATIONS:
Overall Officials: Erwan BORIES, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (3):
- France (2):
  - Institut Paoli-Calmettes, Marseille
  - Hopital Nord, Marseille
- Centre Hospitalier Princesse Grace, Monaco, Monaco

REFERENCES:
- See also: sponsor web site — http://www.institutpaolicalmettes.fr/